CLINICAL TRIAL: NCT02295085
Title: Fernald Community Cohort - 18 Year Observational Study with Bio Banked Blood and Urine Samples
Brief Title: Fernald Community Cohort -18 Year Observational Study
Acronym: FCC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Susan Pinney, Director, Center for Environmental Genetics, Department of Environmental and Public Health Sciences, Program Leader, Cincinnati Cancer Center , UC College of Medicine, University of Cincinnati
Other Study IDs: UC2012-3745; P30ES006096 (NIH)
Record Dates: First submitted 2014-10-29; First posted 2014-11-20 (Estimated); Last update posted 2024-10-26 (Actual); Status verified 2022-03

CONDITIONS: Cancer; Renal Failure; Diabetes; Cardiovascular Disease
Keywords: Cohort, Prospective, Biospecimens
MeSH Terms: conditions — Neoplasms; Renal Insufficiency; Diabetes Mellitus; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 160,000 archived biosamples available, drawn from 1990-2008 (whole Bood, Plasma, Serum, Urine, Buffered Urine), extracted DNA. Breast, Renal & Prostate cancer formalin fixed tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The Fernald Community Cohort consists of the 9782 persons who were enrolled in the Fernald Medical Monitoring Program (FMMP) (1990-2008). The initial comprehensive examination conducted as part of the Fernald Medical Monitoring Program (FMMP) began in the autumn of 1990. The FMMP provided 9,782 initial examinations and 42,775 re-examinations. An extensive computerized database and biospecimen repository was created to provide research resources for future studies. All questionnaire, examination and diagnostic procedure data collected from the FMMP were [coded by certified medical record coders,] double entered with verification into a SAS database on site of the examinations. Cryo-preserved blood and urine samples were collected at enrollment and at various intervals throughout follow-up. At the first examination three 1-ml aliquots of whole blood, plasma, serum, urine and urine with buffer were obtained from each participant (15 aliquots per person) for future analyses. Additional whole blood and serum was obtained in 1996-1997 and 2006-2008. Specimens have been stored in -80 degree freezers; over 160,000 biospecimens are in the archive. Since 1994, the FCC has had an established procedure for sharing data and biospecimens with qualified researchers. Both the policy and application forms can be found at www.eh.uc.edu/fmmp/research.

DETAILED DESCRIPTION:
The Fernald Medical Monitoring Program (FMMP) was designed to provide a comprehensive evaluation of current health and risks for future disease and collect information for subsequent research studies for those who met the enrollment criteria in the FMMP.

Purpose of the FMMP

1. To provide a complete evaluation of current health.
2. To provide a comprehensive evaluation of risk factors for disease, which may develop in the future.
3. To educate on how to reduce the chances of developing disease in the future.
4. Create an epidemiologic database for future studies.

Procedures

1. Consent to participate-The first step in the process was to verbally explain to potential participants the components of the program, the results they would receive, the future use of data and biospecimens. Staff then witnessed their signature on the consent form.
2. Questionnaire- Complete an extensive health questionnaire that was administered each year. Data collected included personal characteristics (age, sex, current address, income, education, marital status, other persons in the home), current and past occupations, family medical history, past addresses and dates. SF-36 (and later the SF-12) health status questionnaire was administered and questions on current diet were asked.
3. History and Physical Examination by physician- A board Certified Physician in Internal Medicine, Occupational Medicine, or Family Practice performed a comprehensive Review of Systems and Physical examination.
4. Laboratory Testing- Blood samples were obtained for a series of screening tests which include complete blood count with differential, blood sugar, thyroid function tests, chemistry liver, kidney and cholesterol profiles. Men age 49-79 were offered a PSA (prostate specific antigen) each year. Urine was collected for urinalysis (occult and microscopic) and a beta2 microglobulin, urine creatine, protein, and microalbumin was completed at the first examination, All Laboratory test results are housed in a SAS database.
5. X-ray Examination- All adults were offered a baseline chest x-ray and offered again at the third through seventh examination cycles. Chest x-ray was offered annually for those with abnormalities. Women 40 years of age or over were offered a screening mammogram each year. The complete narrative of the reports of these procedures has been entered into the SAS database. Findings and recommendations have been coded.
6. Other testing - All adults were offered a baseline electrocardiogram (EKG) and a baseline PFT (pulmonary function test). Those who were age 45 were tested for occult blood in their stool at each examination.
7. Blood and urine samples for research- Blood and urine samples were collected and processed into 15 aliquots (3 whole blood, 3 plasma, 3 serum 3 urine, 3 buffered urine) and frozen in -80 freezers to be used for future epidemiologic studies.

Follow up

At the conclusion of the examination physicians recorded any new medical diagnoses apparent at the time of the examination, as well as diagnostic uncertainties requiring further diagnostic testing. Nurses conducted participant follow up by phone for at least six months on all those needing further testing or treatment by their usual primary care practitioner. New diagnoses recognized through this follow up also are recorded on the medical record. Outside medical records (usually a pathology report) are obtained to validate any new diagnosis of cancer. This same procedure was used at the time of the periodic medical examination offered every three years until 1999. and then every two years until 2008.

Ongoing Questionnaires

Following the initial questionnaire, participants also are asked to complete yearly questionnaire requesting information about new medical problems and recent hospitalizations and surgeries, and 77,638 completed questionnaire from adults have been received by the program. Yearly questionnaire return rates varied by Program year, but in 2008 were 44.8% of the original enrollees. Yearly questionnaire were computer-generated so that participants who missed a past questionnaire are re-issued critical data items from those missed questionnaires, greatly improving total ascertainment on any data item. Continued participation in the program at the time of re-examination fell 23% at the first re-exam for adults and remained at about 50% for each examination since then. (Some participants skip one exam but then return for the next one.) Only 216 participants have withdrawn from the Program and are no longer contacted or followed (except to obtain information when we learn of their death); 184 participants are lost to follow-up. Thus, over 50% of initial participants continued to get semi-annual examinations and we know the location and vital status of 97% of the initial participants.

Follow up time, considering the period under observation to be from the first examination date until the last questionnaire or exam contact, or death, was most program participants, we have 12.5 years of follow-up. Death certificates have been obtained, or an NDI search completed, on most of the 662 participants who have died.

Background of the Fernald Medical Monitoring Program

The Fernald Medical Monitoring Program (FMMP) provided health screenings and health promotion service as the result of a settlement between the US Department of Energy (DOE) and attorneys representing individuals (class members) living or working within five miles of the Feeds Material Processing Center (FMPC), a uranium processing plant in Fernald, Ohio. The lawsuit was based on emotional distress related primarily to the potential for harmful health effects resulting from environmental releases. The settlement also included provisions for supporting epidemiological studies.

This cohort is appropriate to use for studies that are not related to radiation or uranium exposure. Much of the cohort never received uranium exposure beyond the background exposure received by the general population. Extensive uranium dose reconstruction using methods developed by the CDC demonstrate that over 60% of the cohort had such minimal exposure to uranium and radon that their cumulative ionizing radiation exposure was less that 3.2% over lifetime background levels. For the US population, background ionizing radiation exposure is estimated to be 3.6 mSv per year or 288 mSv lifetime (80 Years), but the range of individual exposure estimates is wide, depending primarily on geographic location (1-10 mSv per year). The maximum estimate of yearly exposure beyond background for this 60% sub-cohort is only 5.5 mSv, very small compared to the yearly individual dose variation. Lifetime cumulative exposure from the FMPC for this unexposed sub-group ranges from 0.0 to 0.45 Sv. For the other 40% of the cohort, cumulative lifetime exposure from FMPC ranges (approximately) from 450 mSv (0.45 SV) to 3660 mSv (3.66 Sv).

On January 13, 2013 the Special Master of the Fernald Settlement Fund entered into an agreement to transfer the FMMP database and biospecimen collection to the University of Cincinnati for the purpose of maintaining the database and biospecimen collection for use in epidemiological and genetic research. The Fernald Medical Monitoring Program (FMMP) became the Fernald Community Cohort (FCC).

Strengths of this Program for research

All diagnoses have been assigned ICD-9 codes by a certified medical record coder. All medication information is coded by type of drug using a 4-digit code. The extensive coding of the medical information of this large cohort provides the immediate opportunity to ask specific research questions. For example, all of the 28,518 mammogram reports and the 27,855 chest x-ray reports in the database have been literally coded (coding of phrases) using a list of over 200 3-digit codes, specific to each type of imaging. Exposure or risk factor metrics have been developed from questionnaire information, and are available in the database. For example, we have developed matrix of cumulative cigarette pack-years for all participants, for each year after their year of program enrollment. We also have matrices for family history of each type of cancer for each program participant with number of first degree and total number of blood relatives with that type of cancer.

We have collected family structure information from all participants on several different occasions and through several types of questions (family history at the time of the initial examination, questions about who else lived with you, and questions about offspring on one of the yearly questionnaires).

In each instance, we have recorded names of these relatives and coded each mentioned family member with their FMMP ID, if they are program participants. With each questionnaire we also ask participants of the names of three personal contacts, and record their relationship to the program participants. The FMMP database contains the information needed to create family pedigrees, and note which family members are Program participants.

The extensive information on participants of the FMMP allows for the selection of tailored control groups. Criteria for controls for studies may differ depending on the disease and the lifestyle factor being studied. For example, the FMMP has provided Dr. Marshall Anderson with a set of controls for studies of identified susceptibility genetic variants related to cigarette smoking and lung cancer. For this study, the controls were persons with no first degree relatives with lung cancer, age > 60 years, and with a > 20 pack year cigarette smoking history. Our large cohort and extensive database enabled us to identify more than the needed 200 controls from the group without environmental uranium exposure. We will be conducting a similar control selection for Dr. Daniel Nebert, searching for "highly resistant" persons for his study of susceptibility genes for head and neck cancer but with a > 80 pack year smoking history and no history of any cancer. Persons who meet these criteria are very rare in any population, but we have located 33 controls with these criteria.

The cohort is not racially diversified, which enhances the opportunity for detecting relationships between genomic variation and disease and for discovering biomarker predictors of disease. Since 95% of the cohort is Whit-non-Hispanic, statistical power of genetic studies and precision of data analyses are improved by the lack of racial diversity of this cohort. Although the lack of generalizability to populations with other racial composition is certainly a limitation, the statistical associations found in this population can later be tested in other more racially diverse populations.

The database is an excellent resource for developing methods for data mining, and the potential discovery of new statistical associations will lead to hypothesis generation. The extensive database for this longitudinal cohort provides rich opportunities for data mining, and for developing and testing new method of data mining.

ELIGIBILITY:
Inclusion Criteria:

Lived or worked within five miles of the Feed Material Processing Center (FMPC) for 2 consecutive years between January 1, 1952 and December 18, 1984. The Fernald Community Cohort (N=9782) includes 5294 female and 4489 male participants; 99.5% are Caucasian. The FMMP has conducted 42,775 medical examinations through the end of 2008.

-

Exclusion Criteria:

Worked at the Feeds Material Processing Center (FMPC)

Employed by the US Department of Energy or National Lead of Ohio, Inc. (Plant Contractor)

-

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Community members who lived or worked within the five mile radius of the Fernald Uranium Processing Plant boundary for a least 2 consecutive years between January 1, 1952 and December 18, 1984.
Sampling Method: Non-Probability Sample
Enrollment: 9782 (Actual)
Dates: Start 1990-09; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incident cancer during the period of cohort follow-up | From enrollment to most recent encounter, average of 12 years, range of 1 day to 18 years
  Using information from the medical examinations, medical history, assigned ICD codes and diagnosis verification with pathology reports, cancer outcomes are noted in the database with diagnosis date and method of diagnosis verification.

SECONDARY OUTCOMES:
Incident renal disease during the period of cohort follow-up | From enrollment to most recent encounter, average of 12 years, range of 1 day to 18 years
  Using information from the medical examinations, medical history, laboratory tests of blood serum and urine, and assigned ICD codes, persons with renal disease are noted in the database with diagnosis date and method of diagnosis verification.

OTHER OUTCOMES:
Other incident conditions during the period of cohort followup | From enrollment to most recent encounter, average of 12 years, range of 1 day to 18 years
  Operational definition for diagnosis of medical condition determined by the research conducting the analyses. Operational definition my use information from the medical examinations, medical history, laboratory tests of blood serum and urine, and assigned ICD codes. Persons with that diagnosis are then are noted in the database with diagnosis date and method of diagnosis verification.

CONTACTS AND LOCATIONS:
Overall Officials: Susan M Pinney, PhD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 3. Fitzpatrick S, Nolan RD, Hallam JS, Pinney, SM. Ecological grief in the Fernald Community Cohort: A pilot study. PLOS Mental Health, 1(1): e0000049. https://doi.org/10.1371/journal.pmen.0000049
- [Background] 4. Burcham S, Saul D., Nolan RD., Pinney SM. (2024). Exposure Experiences of Area Residents Near a Chronic Environmental Contamination Site. Ohio Journal of Public Health, 6(1), 1-9. https://doi.org/10.18061/ojph.v6i1.9701
- [Background] Rubinstein J, Pinney SM, Xie C, Wang HS. Association of same-day urinary phenol levels and cardiac electrical alterations: analysis of the Fernald Community Cohort. Environ Health. 2024 Sep 19;23(1):76. doi: 10.1186/s12940-024-01114-x. PMID 39300535
- [Background] Li Y, Xiao X, Li J, Han Y, Cheng C, Fernandes GF, Slewitzke SE, Rosenberg SM, Zhu M, Byun J, Bosse Y, McKay JD, Albanes D, Lam S, Tardon A, Chen C, Bojesen SE, Landi MT, Johansson M, Risch A, Bickeboller H, Wichmann HE, Christiani DC, Rennert G, Arnold SM, Goodman GE, Field JK, Davies MPA, Shete S, Marchand LL, Liu G, Hung RJ, Andrew AS, Kiemeney LA, Sun R, Zienolddiny S, Grankvist K, Johansson M, Caporaso NE, Cox A, Hong YC, Lazarus P, Schabath MB, Aldrich MC, Schwartz AG, Gorlov I, Purrington KS, Yang P, Liu Y, Bailey-Wilson JE, Pinney SM, Mandal D, Willey JC, Gaba C, Brennan P, Xia J, Shen H, Amos CI. Lung Cancer in Ever- and Never-Smokers: Findings from Multi-Population GWAS Studies. Cancer Epidemiol Biomarkers Prev. 2024 Mar 1;33(3):389-399. doi: 10.1158/1055-9965.EPI-23-0613. PMID 38180474
- [Background] Wones R, Pinney SM, Buckholz JM, Deck-Tebbe C, Freyberg R, Pesce A. Medical monitoring: a beneficial remedy for residents living near an environmental hazard site. J Occup Environ Med. 2009 Dec;51(12):1374-83. doi: 10.1097/JOM.0b013e3181c558f1. PMID 19952785
- [Background] Blomkalns AL, Gavrila D, Thomas M, Neltner BS, Blanco VM, Benjamin SB, McCormick ML, Stoll LL, Denning GM, Collins SP, Qin Z, Daugherty A, Cassis LA, Thompson RW, Weiss RM, Lindower PD, Pinney SM, Chatterjee T, Weintraub NL. CD14 directs adventitial macrophage precursor recruitment: role in early abdominal aortic aneurysm formation. J Am Heart Assoc. 2013 Mar 8;2(2):e000065. doi: 10.1161/JAHA.112.000065. PMID 23537804
- [Background] You M, Wang D, Liu P, Vikis H, James M, Lu Y, Wang Y, Wang M, Chen Q, Jia D, Liu Y, Wen W, Yang P, Sun Z, Pinney SM, Zheng W, Shu XO, Long J, Gao YT, Xiang YB, Chow WH, Rothman N, Petersen GM, de Andrade M, Wu Y, Cunningham JM, Wiest JS, Fain PR, Schwartz AG, Girard L, Gazdar A, Gaba C, Rothschild H, Mandal D, Coons T, Lee J, Kupert E, Seminara D, Minna J, Bailey-Wilson JE, Amos CI, Anderson MW. Fine mapping of chromosome 6q23-25 region in familial lung cancer families reveals RGS17 as a likely candidate gene. Clin Cancer Res. 2009 Apr 15;15(8):2666-74. doi: 10.1158/1078-0432.CCR-08-2335. Epub 2009 Apr 7. PMID 19351763
- [Background] Liu P, Vikis HG, Wang D, Lu Y, Wang Y, Schwartz AG, Pinney SM, Yang P, de Andrade M, Petersen GM, Wiest JS, Fain PR, Gazdar A, Gaba C, Rothschild H, Mandal D, Coons T, Lee J, Kupert E, Seminara D, Minna J, Bailey-Wilson JE, Wu X, Spitz MR, Eisen T, Houlston RS, Amos CI, Anderson MW, You M. Familial aggregation of common sequence variants on 15q24-25.1 in lung cancer. J Natl Cancer Inst. 2008 Sep 17;100(18):1326-30. doi: 10.1093/jnci/djn268. Epub 2008 Sep 9. PMID 18780872
- [Background] Liu P, Yang P, Wu X, Vikis HG, Lu Y, Wang Y, Schwartz AG, Pinney SM, de Andrade M, Gazdar A, Gaba C, Mandal D, Lee J, Kupert E, Seminara D, Minna J, Bailey-Wilson JE, Spitz M, Amos CI, Anderson MW, You M. A second genetic variant on chromosome 15q24-25.1 associates with lung cancer. Cancer Res. 2010 Apr 15;70(8):3128-35. doi: 10.1158/0008-5472.CAN-09-3583. PMID 20395203
- [Background] Wagner SE, Burch JB, Bottai M, Pinney SM, Puett R, Porter D, Vena JE, Hebert JR. Hypertension and hematologic parameters in a community near a uranium processing facility. Environ Res. 2010 Nov;110(8):786-97. doi: 10.1016/j.envres.2010.09.004. PMID 20889151
- [Background] Lu-Fritts PY, Kottyan LC, James JA, Xie C, Buckholz JM, Pinney SM, Harley JB. Association of systemic lupus erythematosus with uranium exposure in a community living near a uranium-processing plant: a nested case-control study. Arthritis Rheumatol. 2014 Nov;66(11):3105-12. doi: 10.1002/art.38786. PMID 25103365
- [Background] Fang S, Pinney SM, Bailey-Wilson JE, de Andrade MA, Li Y, Kupert E, You M, Schwartz AG, Yang P, Anderson MW, Amos CI. Ordered subset analysis identifies loci influencing lung cancer risk on chromosomes 6q and 12q. Cancer Epidemiol Biomarkers Prev. 2010 Dec;19(12):3157-66. doi: 10.1158/1055-9965.EPI-10-0792. Epub 2010 Oct 28. PMID 21030603
- [Background] Amos CI, Pinney SM, Li Y, Kupert E, Lee J, de Andrade MA, Yang P, Schwartz AG, Fain PR, Gazdar A, Minna J, Wiest JS, Zeng D, Rothschild H, Mandal D, You M, Coons T, Gaba C, Bailey-Wilson JE, Anderson MW. A susceptibility locus on chromosome 6q greatly increases lung cancer risk among light and never smokers. Cancer Res. 2010 Mar 15;70(6):2359-67. doi: 10.1158/0008-5472.CAN-09-3096. Epub 2010 Mar 9. PMID 20215501
- [Background] Yaghjyan L, Mahoney MC, Succop P, Wones R, Buckholz J, Pinney SM. Relationship between breast cancer risk factors and mammographic breast density in the Fernald Community Cohort. Br J Cancer. 2012 Feb 28;106(5):996-1003. doi: 10.1038/bjc.2012.1. Epub 2012 Jan 26. PMID 22281662
- [Background] Liu P, Vikis HG, Lu Y, Wang Y, Schwartz AG, Pinney SM, Yang P, de Andrade M, Gazdar A, Gaba C, Mandal D, Lee J, Kupert E, Seminara D, Minna J, Bailey-Wilson JE, Amos CI, Anderson MW, You M. Cumulative effect of multiple loci on genetic susceptibility to familial lung cancer. Cancer Epidemiol Biomarkers Prev. 2010 Feb;19(2):517-24. doi: 10.1158/1055-9965.EPI-09-0791. PMID 20142248
- [Background] Christiani DC. Lung cancer genetics: a family affair? Clin Cancer Res. 2009 Apr 15;15(8):2581-2. doi: 10.1158/1078-0432.CCR-09-0003. Epub 2009 Apr 7. PMID 19351746
- [Background] Xiong D, Wang Y, Kupert E, Simpson C, Pinney SM, Gaba CR, Mandal D, Schwartz AG, Yang P, de Andrade M, Pikielny C, Byun J, Li Y, Stambolian D, Spitz MR, Liu Y, Amos CI, Bailey-Wilson JE, Anderson M, You M. A recurrent mutation in PARK2 is associated with familial lung cancer. Am J Hum Genet. 2015 Feb 5;96(2):301-8. doi: 10.1016/j.ajhg.2014.12.016. Epub 2015 Jan 29. PMID 25640678
- [Background] Yang S, Pinney SM, Mallick P, Ho SM, Bracken B, Wu T. Impact of Oxidative Stress Biomarkers and Carboxymethyllysine (an Advanced Glycation End Product) on Prostate Cancer: A Prospective Study. Clin Genitourin Cancer. 2015 Oct;13(5):e347-51. doi: 10.1016/j.clgc.2015.04.004. Epub 2015 Apr 18. PMID 25972296
- [Background] Pinney SM, Biro FM. Letter to the editor re Morollo-Frosh "Communicating results in post-Belmont era biomonitoring studies". Environ Res. 2015 Oct;142:756. doi: 10.1016/j.envres.2015.05.024. Epub 2015 Jun 12. No abstract available. PMID 26076818
- [Background] Liu Y, Kheradmand F, Davis CF, Scheurer ME, Wheeler D, Tsavachidis S, Armstrong G, Simpson C, Mandal D, Kupert E, Anderson M, You M, Xiong D, Pikielny C, Schwartz AG, Bailey-Wilson J, Gaba C, De Andrade M, Yang P, Pinney SM; Genetic Epidemiology of Lung Cancer Consortium; Amos CI, Spitz MR. Focused Analysis of Exome Sequencing Data for Rare Germline Mutations in Familial and Sporadic Lung Cancer. J Thorac Oncol. 2016 Jan;11(1):52-61. doi: 10.1016/j.jtho.2015.09.015. PMID 26762739
- [Background] Martin AT, Pinney SM, Xie C, Herrick RL, Bai Y, Buckholz J, Martin VT. Headache Disorders May Be a Risk Factor for the Development of New Onset Hypothyroidism. Headache. 2017 Jan;57(1):21-30. doi: 10.1111/head.12943. Epub 2016 Sep 27. PMID 27676320
- [Background] Herrick RL, Buckholz J, Biro FM, Calafat AM, Ye X, Xie C, Pinney SM. Polyfluoroalkyl substance exposure in the Mid-Ohio River Valley, 1991-2012. Environ Pollut. 2017 Sep;228:50-60. doi: 10.1016/j.envpol.2017.04.092. Epub 2017 May 13. PMID 28505513
- [Background] Giannini CM, Herrick RL, Buckholz JM, Daniels AR, Biro FM, Pinney SM. Comprehension and perceptions of study participants upon receiving perfluoroalkyl substance exposure biomarker results. Int J Hyg Environ Health. 2018 Aug;221(7):1040-1046. doi: 10.1016/j.ijheh.2018.07.005. Epub 2018 Jul 17. PMID 30025914
- [Background] Greene AD, Kendziorski JA, Buckholz JM, Niu L, Xie C, Pinney SM, Burns KA. Elevated serum chemokines are independently associated with both endometriosis and uranium exposure. Reprod Toxicol. 2019 Mar;84:26-31. doi: 10.1016/j.reprotox.2018.12.006. Epub 2018 Dec 21. PMID 30579999
- [Background] Blake BE, Pinney SM, Hines EP, Fenton SE, Ferguson KK. Associations between longitudinal serum perfluoroalkyl substance (PFAS) levels and measures of thyroid hormone, kidney function, and body mass index in the Fernald Community Cohort. Environ Pollut. 2018 Nov;242(Pt A):894-904. doi: 10.1016/j.envpol.2018.07.042. Epub 2018 Jul 17. PMID 30373035
- [Background] Byun J, Schwartz AG, Lusk C, Wenzlaff AS, de Andrade M, Mandal D, Gaba C, Yang P, You M, Kupert EY, Anderson MW, Han Y, Li Y, Qian D, Stilp A, Laurie C, Nelson S, Zheng W, Hung RJ, Gaborieau V, Mckay J, Brennan P, Caporaso NE, Landi MT, Wu X, McLaughlin JR, Brhane Y, Bosse Y, Pinney SM, Bailey-Wilson JE, Amos CI. Genome-wide association study of familial lung cancer. Carcinogenesis. 2018 Sep 21;39(9):1135-1140. doi: 10.1093/carcin/bgy080. PMID 29924316
- [Background] Liu Y, Lusk CM, Cho MH, Silverman EK, Qiao D, Zhang R, Scheurer ME, Kheradmand F, Wheeler DA, Tsavachidis S, Armstrong G, Zhu D, Wistuba II, Chow CB, Behrens C, Pikielny CW, Neslund-Dudas C, Pinney SM, Anderson M, Kupert E, Bailey-Wilson J, Gaba C, Mandal D, You M, de Andrade M, Yang P, Field JK, Liloglou T, Davies M, Lissowska J, Swiatkowska B, Zaridze D, Mukeriya A, Janout V, Holcatova I, Mates D, Milosavljevic S, Scelo G, Brennan P, McKay J, Liu G, Hung RJ, Christiani DC, Schwartz AG, Amos CI, Spitz MR. Rare Variants in Known Susceptibility Loci and Their Contribution to Risk of Lung Cancer. J Thorac Oncol. 2018 Oct;13(10):1483-1495. doi: 10.1016/j.jtho.2018.06.016. Epub 2018 Jul 4. PMID 29981437
- [Background] Musolf AM, Moiz BA, Sun H, Pikielny CW, Bosse Y, Mandal D, de Andrade M, Gaba C, Yang P, Li Y, You M, Govindan R, Wilson RK, Kupert EY, Anderson MW, Schwartz AG, Pinney SM, Amos CI, Bailey-Wilson JE. Whole Exome Sequencing of Highly Aggregated Lung Cancer Families Reveals Linked Loci for Increased Cancer Risk on Chromosomes 12q, 7p, and 4q. Cancer Epidemiol Biomarkers Prev. 2020 Feb;29(2):434-442. doi: 10.1158/1055-9965.EPI-19-0887. Epub 2019 Dec 11. PMID 31826912
- [Background] Liu Y, Xia J, McKay J, Tsavachidis S, Xiao X, Spitz MR, Cheng C, Byun J, Hong W, Li Y, Zhu D, Song Z, Rosenberg SM, Scheurer ME, Kheradmand F, Pikielny CW, Lusk CM, Schwartz AG, Wistuba II, Cho MH, Silverman EK, Bailey-Wilson J, Pinney SM, Anderson M, Kupert E, Gaba C, Mandal D, You M, de Andrade M, Yang P, Liloglou T, Davies MPA, Lissowska J, Swiatkowska B, Zaridze D, Mukeria A, Janout V, Holcatova I, Mates D, Stojsic J, Scelo G, Brennan P, Liu G, Field JK, Hung RJ, Christiani DC, Amos CI. Rare deleterious germline variants and risk of lung cancer. NPJ Precis Oncol. 2021 Feb 16;5(1):12. doi: 10.1038/s41698-021-00146-7. PMID 33594163
- [Background] Musolf AM, Simpson CL, Moiz BA, Pikielny CW, Middlebrooks CD, Mandal D, de Andrade M, Cole MD, Gaba C, Yang P, You M, Li Y, Kupert EY, Anderson MW, Schwartz AG, Pinney SM, Amos CI, Bailey-Wilson JE. Genetic Variation and Recurrent Haplotypes on Chromosome 6q23-25 Risk Locus in Familial Lung Cancer. Cancer Res. 2021 Jun 15;81(12):3162-3173. doi: 10.1158/0008-5472.CAN-20-3196. Epub 2021 Apr 14. PMID 33853833
- See also: website — https://med.uc.edu/depart/eh/research/projects/fcc/home